CLINICAL TRIAL: NCT02697825
Title: Correlation Between Intraocular Pressure and Optic Nerve Sheath Diameter
Brief Title: Intraocular Pressure Versus Optic Nerve Sheath Diameter
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Rajiv Gandhi Cancer Institute & Research Center, India (Other)
Responsible Party: Principal Investigator, Dr. Nitesh Goel, Doctor Nitesh Goel, Consultant Anaesthesia, Rajiv Gandhi Cancer Institute & Research Center, India
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: RajivGCIRC1
Record Dates: First submitted 2016-02-20; First posted 2016-03-03 (Estimated); Last update posted 2016-03-03 (Estimated); Status verified 2016-02

CONDITIONS: Intraocular Pressure; Optic Nerve Sheath Diameter
MeSH Terms: interventions — Intraocular Pressure; High-Energy Shock Waves

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- changes in eye (Other): Changes in both intraocular pressure and optic nerve sheath diameter will be correlated in robotic surgeries to find out any statistical relation existing between two.
  Interventions: Procedure: Schiotz tonometer for Intraocular Pressure

INTERVENTIONS:
Procedure: Schiotz tonometer for Intraocular Pressure — Both Values will be corelated
  Other Names: Ultrasound for Optic nerve sheath diameter

SUMMARY:
This study involves observing and comparing Intraocular Pressure and Optic Nerve Sheath Diameter in steep trendelenburg position. Both observations will be done in same patient over the surgical duration.

DETAILED DESCRIPTION:
Steep trendelenburg position is required for various robotic surgical procedures like hysterectomy, radical prostatectomy etc. Both Intraocular Pressure and Optic Nerve Sheath Diameter are found to get increased while in this position.

Intraocular Pressure will be measured by schiotz tonometer over an hourly interval whereas Optic nerve sheath diameter will be measured with use of ultrasound using a probe of 7.5 Mega hertz. Both values will be measured in both the eyes and will be compared statistically to find any correlation which may exist between the two.

ELIGIBILITY:
Inclusion Criteria:

* robotic surgeries
* surgical duration upto 4 hours
* american society of anaesthesiologists 1 to 3

Exclusion Criteria:

* any history of opthalmic intervention
* patient suffering from glaucoma
* patients taking any diuretics for cardiac problems

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2015-09; Primary Completion 2016-03 (Estimated); Study Completion 2016-04 (Estimated)

PRIMARY OUTCOMES:
correlation between rise of intraocular pressure and optic nerve sheath diameter | 9 months
  Intraocular pressure will be measured using schiotz tonometer whereas optic nerve sheath diameter will be assessed using ultrasound in same patient at same intervals. This will give us both the values of intraocular pressure and optic nerve sheath diameter at same time which as per previous studies increases and are statistically significant. After compilation of results it will be analyzed that whether both values increases in a correlated manner or not which will give us our results that whether increase of one value can tell the increase of other value.

CONTACTS AND LOCATIONS:
Overall Officials: Nitesh Goel, MBBS,DA, DNB, Principal Investigator — Rajiv Gandhi Cancer Institute & Research Centre
Locations (1):
- Rajiv Gandhi Cancer Institute & Research Centre, New Delhi, National Capital Territory of Delhi, India

IPD SHARING:
Plan to Share IPD: Undecided
It will be decide only after the completion of study